CLINICAL TRIAL: NCT01635647
Title: A Phase 1/2b Double Blind Randomised Controlled Trial of the Efficacy, Safety and Immunogenicity of Heterologous Prime-boost Immunisation With the Candidate Malaria Vaccines ChAd63 ME-TRAP and MVA ME-TRAP in 5-17 Month Old Burkinabe Infants and Children
Brief Title: A Phase 1/2b Study of an Investigational Malaria Vaccination Strategy in 5-17 Month Old Infants and Children in Burkina Faso
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAC050
Record Dates: First submitted 2012-07-03; First posted 2012-07-09 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ChAd63 ME-TRAP and MVA ME-TRAP (Active Comparator): ChAd63 ME-TRAP / MVA ME-TRAP heterologous prime-boost immunisation
  Interventions: Biological: ChAd63 ME-TRAP and MVA ME-TRAP
- Rabies vaccine (Placebo Comparator): 2 x 2.5IU Verorab
  Interventions: Biological: Rabies vaccine

INTERVENTIONS:
Biological: ChAd63 ME-TRAP and MVA ME-TRAP — ChAd63 ME-TRAP: 5 x 10^10vp MVA ME-TRAP: 1 x 10^8 pfu heterologous prime-boost immunisation
  Arms: ChAd63 ME-TRAP and MVA ME-TRAP
Biological: Rabies vaccine — Two doses eight weeks apart into anterolateral thigh. 2 x 2.5IU Verorab
  Arms: Rabies vaccine

SUMMARY:
Prime boost vaccination with ChAd63 ME-TRAP followed eight weeks later with MVA ME-TRAP shows efficacy against malaria infection when tested in UK volunteers using sporozoite challenge experiments. It is a leading candidate vaccination strategy against malaria. In the field, Phase I studies have been conducted in adults in Kenya and The Gambia and children and infants in The Gambia. The vaccination strategy appears safe and well tolerated in these populations, and also shows impressive immunogenicity, not significantly different to that seen in the UK trials where efficacy was shown. In particular, recent data from The Gambia shows excellent safety and immunogenicity in infants in malaria endemic areas, who would be the ones to benefit most from such a vaccine against malaria. With this clinical development as background, the investigators now propose to evaluate efficacy against natural malaria infection in this important target group for an effective malaria vaccine, that is, 5-17 month infants and children living in malaria endemic areas. The proposed study area, Banfora, Burkina Faso, is highly endemic for Plasmodium falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infant/child aged 5-17 months at the time of first study vaccination
2. Informed consent of parent/guardian
3. Infant / child and parent/guardian resident in the study area villages and anticipated to be available for vaccination and follow-up

Exclusion Criteria:

* Clinically significant skin disorder (psoriasis, contact dermatitis etc.), immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness.
* Weight-for-age Z score of less than -3 or other clinical signs of malnutrition
* History of allergic reaction, significant IgE-mediated event, or anaphylaxis to immunisation
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, e.g. egg products, Kathon, neomycin, beta-propiolactone.
* Haemoglobin less than 8.0 g/dL, where judged to be clinically significant in the opinion of the investigator
* Serum Creatinine concentration greater than 70 µmol/L, where judged to be clinically significant in the opinion of the investigator
* Serum ALT concentration greater than 45 U/L, where judged to be clinically significant in the opinion of the investigator
* Blood transfusion within one month of enrolment
* Previous vaccination with experimental malaria vaccines.
* Administration of any other vaccine or immunoglobulin less than one week before vaccination with any study vaccine.
* Current participation in another clinical trial, or within 12 weeks of this study.
* Any other finding which in the opinion of the investigators would increase the risk of an adverse outcome from participation in the trial or result in incomplete or poor quality data
* Known maternal HIV infection (No testing will be done by the study team)
* Immunosuppressive therapy (steroids, immune modulators or immune suppressors) within 3 months prior recruitment. (For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)

Ages: 5 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 730 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Time to first episode of malaria meeting the primary case definition of clinical malaria episode | 6 months

SECONDARY OUTCOMES:
Duration of Protective efficacy against clinical malaria | 12 and 24 months
  To assess the protective efficacy against clinical malaria of ChAd63 ME-TRAP / MVA ME-TRAP prime-boost immunisation, in 5-17 month old infants and children living in a malaria-endemic area, for 12 and 24* months after the last vaccination.
Efficacy against asymptomatic P. falciparum infection | 6, 12 and 24 months
  To assess the protective efficacy against asymptomatic P. falciparum infection of ChAd63 ME-TRAP / MVA ME-TRAP prime-boost immunisation, in 5-17 month old infants and children living in a malaria-endemic area, 6, 12 and 24* months after the last vaccination
Efficacy against secondary case definitions of clinical malaria | 6, 12 and 24 months
  To assess the protective efficacy against secondary case definitions of clinical malaria of ChAd63 ME-TRAP / MVA ME-TRAP prime-boost immunisation, in 5-17 month old infants and children living in a malaria-endemic area, for 6, 12 and 24 months after the last vaccination
Safety Objective | 6, 12 and 24 months
  To assess the safety and reactogenicity of ChAd63 ME-TRAP / MVA ME-TRAP heterologous prime-boost immunisation, in 5-17 month old infants and children living in a malaria-endemic area, for 6, 12 and 24 months after the last vaccination.
Immunogenicity Objectives | 24 months
  * To assess the immunogenicity of ChAd63 ME-TRAP / MVA ME- TRAP heterologous prime-boost immunisation, in 5-17 month old infants and children living in a malaria-endemic area.
  * To explore the immunologic correlates of protective efficacy of ChAd63 ME-TRAP / MVA ME-TRAP prime-boost immunisation, in 5-17 month old infants and children living in a malaria-endemic area.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical Vaccinology and 1. Centre National de Recherche et de Formation sur le Paludisme (CNRFP)/ Unité de Recherche Clinique de Banfora (URC-B), Ouagadougou, Burkina Faso

REFERENCES:
- [Derived] Morter R, Tiono AB, Nebie I, Hague O, Ouedraogo A, Diarra A, Viebig NK, Hill AVS, Ewer KJ, Sirima SB. Impact of exposure to malaria and nutritional status on responses to the experimental malaria vaccine ChAd63 MVA ME-TRAP in 5-17 month-old children in Burkina Faso. Front Immunol. 2022 Dec 2;13:1058227. doi: 10.3389/fimmu.2022.1058227. eCollection 2022. PMID 36532031
- [Derived] Tiono AB, Nebie I, Anagnostou N, Coulibaly AS, Bowyer G, Lam E, Bougouma EC, Ouedraogo A, Yaro JBB, Barry A, Roberts R, Rampling T, Bliss C, Hodgson S, Lawrie A, Ouedraogo A, Imoukhuede EB, Ewer KJ, Viebig NK, Diarra A, Leroy O, Bejon P, Hill AVS, Sirima SB. First field efficacy trial of the ChAd63 MVA ME-TRAP vectored malaria vaccine candidate in 5-17 months old infants and children. PLoS One. 2018 Dec 12;13(12):e0208328. doi: 10.1371/journal.pone.0208328. eCollection 2018. PMID 30540808